CLINICAL TRIAL: NCT06501456
Title: Evaluation of the Relationship Between Non-attendance to Appointments and Adherence to Medical Indications, in Adult Patients, With Type 2 Diabetes Mellitus, During the COVID-19 Pandemic: Cross-sectional Studio.
Brief Title: Evaluation of the Relationship Between Missed Appointments and Adherence to Medical Indications
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, Principal investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 5595
Record Dates: First submitted 2021-05-27; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: No-Show Patients; Therapeutic Adherence and Compliance; Type 2 Diabetes Mellitus; COVID-19
Keywords: No Show Patients; Patient Compliance; Type 2 diabetes mellitus; COVID-19
MeSH Terms: conditions — No-Show Patients; Treatment Adherence and Compliance; Diabetes Mellitus, Type 2; COVID-19; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will conduct a cross-sectional study involving adults with type 2 diabetes mellitus. Our primary objective is to evaluate the association between nonattendance and participants' adherence to both pharmacological and non-pharmacological medical recommendations, as well as COVID-19 prevention measures. Additionally, we will assess the adherence rates to these medical recommendations, COVID-19 prevention protocols, and the recommended health care practices and controls for patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Non-attendance at outpatient visits and lack of adherence to medical recommendations are prevalent issues that negatively impact the health care system. While tools exist to assess pharmacological adherence, evaluating adherence to non-pharmacological recommendations remains challenging. Some studies suggest using nonattendance as an objective and easily measurable marker of adherence.

The aim of this study is to evaluate the association between nonattendance and adherence to medical recommendations in adults with type 2 diabetes mellitus.

We will conduct a cross-sectional study involving adults with type 2 diabetes mellitus. We will evaluate the association between participants' nonattendance and their adherence to both pharmacological and non-pharmacological medical recommendations, as well as COVID-19 prevention measures. Additionally, we will assess the adherence rates to these recommendations, COVID-19 prevention measures, and the recommended health care practices and controls for patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old), affiliated with the medical insurance of the Hospital Italiano de Buenos Aires for at least two years.
* Patients with a diagnosis of type 2 diabetes mellitus at least 2 years before the date of entry to the study Will be included.

Exclusion Criteria:

* Refusal to participate or to the informed consent process.
* Difficulties with language or comprehension (includes pathologies that alter the understanding of the indications or compliance with them (dementia, encephalopathy, intellectual disability, psychiatric disorders).
* Recent hospitalization (the month before the phone call).
* Medical follow-up outside of Hospital Italiano de Buenos Aires.
* Work as health personnel.
* Communication failure (wrong phone number or no response to 3 calls on different days and times)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosis of type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Association between non-attendance to scheduled outpatient shifts and adherence to doctor's instructions in adult patients | 2020 - 2021
  Measured the association between absenteeism from outpatient visits and adherence to medical indications in adults with type 2 diabetes mellitus.

SECONDARY OUTCOMES:
Adherence of patients with type 2 diabetes mellitus to medical indications during the pandemic | July 2020
  Report the adherence of patients with type 2 diabetes mellitus to medical indications during the pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Javier Nicolás Giunta, MD, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zeleke Negera G, Charles Epiphanio D. Prevalence and Predictors of Nonadherence to Diet and Physical Activity Recommendations among Type 2 Diabetes Patients in Southwest Ethiopia: A Cross-Sectional Study. Int J Endocrinol. 2020 Feb 28;2020:1512376. doi: 10.1155/2020/1512376. eCollection 2020. PMID 32190048
- [Result] Brewster S, Bartholomew J, Holt RIG, Price H. Non-attendance at diabetes outpatient appointments: a systematic review. Diabet Med. 2020 Sep;37(9):1427-1442. doi: 10.1111/dme.14241. Epub 2020 Feb 3. PMID 31968127
- [Result] American Diabetes Association. 5. Facilitating Behavior Change and Well-being to Improve Health Outcomes: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S48-S65. doi: 10.2337/dc20-S005. PMID 31862748
- [Result] Sun CA, Taylor K, Levin S, Renda SM, Han HR. Factors associated with missed appointments by adults with type 2 diabetes mellitus: a systematic review. BMJ Open Diabetes Res Care. 2021 Mar;9(1):e001819. doi: 10.1136/bmjdrc-2020-001819. PMID 33674280
- [Result] Lee RRS, Samsudin MI, Thirumoorthy T, Low LL, Kwan YH. Factors affecting follow-up non-attendance in patients with Type 2 diabetes mellitus and hypertension: a systematic review. Singapore Med J. 2019 May;60(5):216-223. doi: 10.11622/smedj.2019042. PMID 31187148
- [Result] Pourhabibi N, Mohebbi B, Sadeghi R, Shakibazadeh E, Sanjari M, Tol A, Yaseri M. Determinants of Poor Treatment Adherence among Patients with Type 2 Diabetes and Limited Health Literacy: A Scoping Review. J Diabetes Res. 2022 Jul 4;2022:2980250. doi: 10.1155/2022/2980250. eCollection 2022. PMID 35832786
- [Result] Giunta D, Briatore A, Baum A, Luna D, Waisman G, de Quiros FG. Factors associated with nonattendance at clinical medicine scheduled outpatient appointments in a university general hospital. Patient Prefer Adherence. 2013 Nov 8;7:1163-70. doi: 10.2147/PPA.S51841. eCollection 2013. PMID 24235820
- [Result] Giunta DH, Alonso Serena M, Luna D, Peroni ML, Sanchez Thomas D, Binder F, Blugerman GA, Fuentes N, Elizondo CM, Gonzalez Bernaldo de Quiros F. Association between non-attendance to outpatient clinics and emergency department consultations, hospitalizations and mortality in a Health Maintenance Organization. Int J Health Plann Manage. 2020 Sep;35(5):1140-1156. doi: 10.1002/hpm.3021. Epub 2020 Jul 9. PMID 32648278
- [Result] Giunta DH, Alonso Serena M. Nonattendance rates of scheduled outpatient appointments in a university general hospital. Int J Health Plann Manage. 2019 Oct;34(4):1377-1385. doi: 10.1002/hpm.2797. Epub 2019 May 7. PMID 31062463
- See also: INDEC Argentina — https://www.indec.gob.ar/ftp/cuadros/poblacion/cuestionario_basico_2010.pdf